CLINICAL TRIAL: NCT01257048
Title: An Open, Randomised, Parallel Group Multi-centre, Methodology Study, Evaluating the Sensitivity of Oxygen-Enhanced Magnetic Resonance Imaging (OE-MRI) in Detecting and Comparing Response to 8 Weeks Treatment With Budesonide/Formoterol Turbuhaler® (320/9 µg Bid) and Formoterol Turbuhaler® (9 µg Bid) in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Evaluation of an Oxygen Enhanced Magnetic Resonance Imaging Method on Patients With Chronic Obstructive Pulmonary Disease During 8 Weeks Treatment With Either Symbicort Turbuhaler or Oxis Turbuhaler
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D6256M00046; 2010-023751
Record Dates: First submitted 2010-12-03; First posted 2010-12-09 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: COPD Method Evaluation; Chronic Obstructive Pulmonary Disease Method Evaluation
Keywords: Oxygen enhanced magnetic resonance imaging; chronic obstructive pulmonary disease; method evaluation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide

ARMS (2):
- 1 (Placebo Comparator): Single Dose evaluation placebo (V5)
  Interventions: Drug: Formoterol Turbuhaler
- 2 (Active Comparator): Single Dose evaluation formoterol (V5)
  Interventions: Drug: Budesonide/Formoterol Turbuhaler; Drug: Formoterol Turbuhaler

INTERVENTIONS:
Drug: Formoterol Turbuhaler — 9 microgram on visit 5 single dose
  Arms: 1
Drug: Budesonide/Formoterol Turbuhaler — 320/9 microgram twice daily during 8 weeks
  Arms: 2
Drug: Formoterol Turbuhaler — 9 microgram twice daily during 8 weeks
  Arms: 2

SUMMARY:
The main purpose of this study is to evaluate the sensitivity of a new oxygen enhanced magnetic resonance imaging (OE-MRI) method in detecting changes in the lungs of patients with moderate to severe chronic obstructive pulmonary disease (COPD) following treatment with either Oxis Turbuhaler or Symbicort Turbuhaler.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 40 years
* Male and female
* Clinical diagnosis of moderate to severe COPD according GOLD guidelines
* Current or ex smoker with a smoking history equivalent to at least 20 cigarettes smoked per day for 10 years
* A Modified Medical Research Council (MMRC) dyspnoea scale score of ≥2.
* FEV1/FVC < 0.7 (post-bronchodilator)
* FEV1 > 40 % PN and < 70 % PN (post-bronchodilator)

Clinical Study Protocol Local Amendment affects UK:

- FEV1 > 30 % PN and < 80 % PN (post-bronchodilator)

Exclusion Criteria:

* Current diagnosis of asthma according to GINA guidelines
* Pregnancy, breast-feeding or planned pregnancy during the study. Fertile women not using acceptable contraceptive measures as judged by the investigator
* Significant upper or lower respiratory tract infection not fully recovered in the 4 weeks prior to visit 1
* Participation in or scheduled for an intensive COPD rehabilitation program
* Claustrophobia, pacemaker, clips within the brain, previous brain or heart surgery, history of metal in the eye or other MRI contraindication such as obesity or inability to stay in the supine position for 60 minutes

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Oxygen enhanced MRI V4 | Visit 4
  Oxygen enhanced magnetic resonance imaging (OE-MRI) parameters
Oxygen enhanced MRI V5 | Visit 5
  Oxygen enhanced MRI parameters
Oxygen enhanced MRI V7 | Visit 7
  Oxygen enhanced MRI parameters

SECONDARY OUTCOMES:
Transferability of OE-MRI technique | 10 months
  Transferability of OE-MRI technique to a second centre
OE-MRI variables | patients will fill in a patient diary at home between visit 2 and 7
  Relationship with OE-MRI variables and change in lung function
Impulse oscillometry parameters V2 | Visit 2
  Impulse oscillometry parameters
Impulse oscillometry parameters V4 | Visit 4
  Impulse oscillometry parameters
Impulse oscillometry parameters V5 | Visit 5
  Impulse oscillometry parameters
Impulse oscillometry parameters V7 | Visit 7
  Impulse oscillometry parameters

CONTACTS AND LOCATIONS:
Locations (2):
- Research Site, Lund, Sweden
- Research Site, Manchester, United Kingdom